CLINICAL TRIAL: NCT03945955
Title: Melatonin Supplementation and Oxidative DNA Damage Repair Capacity Among Night Shift Workers: a Randomized Placebo-controlled Trial
Brief Title: Melatonin and DNA Damage Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Parveen Bhatti, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H19-00780
Record Dates: First submitted 2019-04-30; First posted 2019-05-10 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Sleep Quality; DNA Damage Repair Deficiency; Oxidative Stress
Keywords: Melatonin, Sleep quality, DNA Damage, Lipid peroxidation, Nightshift worker
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental)
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Participants will be randomized into two groups (Group A and Group B). Group A will initially be treated with 3 mg melatonin supplements over a 4-week period while Group B will initially receive placebo supplements over a 4-week period. After a 4-week washout period, Group A will receive placebo supplements while Group B will receive 3 mg melatonin supplements.
  Arms: Melatonin
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This research aims to determine if melatonin supplementation, through improvements in sleep quality, increases the ability to repair oxidative DNA damage and reduce lipid peroxidation levels among nightshift workers.

DETAILED DESCRIPTION:
Administering a 3 mg melatonin supplement to nightshift workers prior to day sleep may significantly improve their oxidative DNA damage repair capacity and reduce the occurrence of lipid peroxidation [measured as increased excretion of urinary 8-hydroxydeoxyguanosine (8-OH-dG) and decreased excretion of urinary 8-isoprostane, respectively] through improvements in sleep quality (measured via actigraphy) and melatonin's direct antioxidative properties.

ELIGIBILITY:
Eligibility criteria included: 1) living and working in the Greater Vancouver area; 2) being between the ages of 18 and 50; 3) having a body mass index (BMI) between 18.5 and 30 kg/m2; 4) working at least two consecutive night shifts per week (≥7 hours per night ending no earlier than 06:00) for at least six months; 5) sleeping, on average, six hours during day sleep periods; 6) not currently using marijuana or illicit drugs; 7) no personal history of sleep disorders, hormone disorders, seizure disorders, or chronic medical conditions (e.g., cancer, diabetes, kidney disease, liver disease, asthma, cardiovascular disease, and infectious disease); 8) not currently pregnant or currently breast feeding; 9) no trans-meridian travel within fours weeks of data collection; and 10) not currently using melatonin supplements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Oxidative DNA damage repair capacity | During day sleep and during night work at baseline and one month
  Measured as urinary concentration of 8-hydroxydeoxyguanosine (ng/mg-Creatinine) between baseline and one month as measured using liquid chromatography tandem mass spectrometry
Sleep duration | During day sleep at baseline and one month
  Measured sleep duration (total minutes asleep) using wrist-based actigraphy device
Karolinska Sleepiness Scale | During night shift work at baseline and one month
  Self-reported level of sleepiness on 9 point scale

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Research Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhatti P, Mirick DK, Randolph TW, Gong J, Buchanan DT, Zhang JJ, Davis S. Oxidative DNA damage during night shift work. Occup Environ Med. 2017 Sep;74(9):680-683. doi: 10.1136/oemed-2017-104414. Epub 2017 Jun 26. PMID 28652381
- [Result] Mirick DK, Bhatti P, Chen C, Nordt F, Stanczyk FZ, Davis S. Night shift work and levels of 6-sulfatoxymelatonin and cortisol in men. Cancer Epidemiol Biomarkers Prev. 2013 Jun;22(6):1079-87. doi: 10.1158/1055-9965.EPI-12-1377. Epub 2013 Apr 5. PMID 23563887
- [Result] Bhatti P, Mirick DK, Davis S. The impact of chronotype on melatonin levels among shift workers. Occup Environ Med. 2014 Mar;71(3):195-200. doi: 10.1136/oemed-2013-101730. Epub 2014 Jan 7. PMID 24399070